CLINICAL TRIAL: NCT03604302
Title: Identification of Essential Areas of the Brain in Pre-Operative Brain Tumor Patients Using BOLD fMRI and Independent Physiological Parameters
Brief Title: Evaluation of Preoperative Functional Magnetic Resonance Imaging (fMRI) in Patients With Brain Tumors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-331
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Brain Tumor
Keywords: Functional Magnetic Resonance Imaging (fMRI); 18-331
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Functional Magnetic Resonance Imaging (fMRI) (Experimental): The interventions for this study are non-invasive. For patients, routine pre-operative MRI that includes task based fMRI and perfusion data acquisition will be performed on a 3T scanner. Patients who participate in this study, will have approximately 5 minutes added to their scan time for the below described breath holding fMRI (BH fMRI) paradigm, which will be done for research purposes. For healthy volunteers, participation will involve having a high resolution anatomical MRI done with the same paradigms which patients will have, listed below. the total scanner time will be approximately 25 minutes, and the scan will not be billed to the healthy volunteer.
  Interventions: Device: fMRI Paradigms

INTERVENTIONS:
Device: fMRI Paradigms — T2*-weighted images will be acquired with a single-shot gradient echo echo-planar imaging (EPI) sequence in the axial orientation (TR=2500ms, TE=30ms, FA=80°, slice thickness=4 mm, FOV= 240mm2, matrix=64×64) covering the whole brain.

SUMMARY:
The purpose of this study is to test the accuracy of using an imaging technique called breath-holding functional magnetic resonance imaging (BH fMRI) in addition to the standard imaging test described above. This study will allow the researchers to find out whether using BH fMRI in combination with the standard approach is the same as, better, or worse than the standard approach used alone.

ELIGIBILITY:
Inclusion Criteria:

Health Volunteers

* Volunteers between the ages of 18 and 80 years
* Volunteers must be able to perform the language paradigms on cue while inside the scanner Patients
* Patients between the ages of 18 and 80 years
* Patients must be able to perform the language paradigms on cue while inside the scanner
* Women of child bearing potential must have a negative pregnancy test prior to the study intervention (Serum or Urine)
* Patients diagnosed with primary glial neoplasm, meningioma and metastasis (from prior histology) or must be suspected to have primary glial neoplasm, meningioma and metastasis on imaging (to be confirmed by post-operative histology).
* Patient"s location of the tumor must involve the expected location of Broca"s area (left pars opercularis and/or pars triangularis), or the expected location of the primary motor area (the pre-central gyrus). This determination will be made on the basis of a pre-operative MRI by a fellowship-trained Neuroradiologist

Exclusion Criteria:

Healthy Volunteers

* Volunteers who are unable to comply or complete MRI exams as per the site"s standards. (e.g.: claustrophobia, high levels of anxiety, pacemaker etc.)

  o MSK site only - see Appendix 2
* Volunteers who are unable to perform the language paradigms on cue while inside the scanner (due to weakness, deafness, inability to understand or follow instructions etc.)
* Volunteers with a history of neurological disorders, psychiatric disorders or cancer Female volunteers who are pregnant or nursing.
* Volunteers who have MRI safe pacemakers.
* Volunteers from the vulnerable population, as defined by 45 CFR 46
* Volunteers who are unable to perform the breath hold task during practice sessions Patients
* Patients who are unable to comply or complete MRI exams as per the site"s standards. (e.g.: claustrophobia, high levels of anxiety, pacemaker etc.)

  °MSK site only - see Appendix 2
* Patients who have MRI safe pacemakers.
* Patient who are unable to perform the language paradigms on cue while inside the scanner (due to weakness, deafness, inability to understand or follow instructions etc.)
* Female patients who are pregnant or nursing.
* Patients from the vulnerable population, as defined by 45 CFR 46
* Patients who are unable to perform the breath hold task during practice sessions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients that have false negative results | 2 years
  The primary objective is to examine if the false negative results of BOLD fMRI adjacent to brain tumors can be compensated for by measurements of BH-MRI and subsequent calibration of the BOLD response. We will have two sets of data: 1) the data obtained using routine techniques to analyze the BOLD fMRI data; and 2) the data obtained where the BOLD fMRI data was analyzed incorporating BH data. Every data point obtained in 1) will have a corresponding data point using 2), the BH MRI data, to adjust the BOLD fMRI analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Holodny, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm